CLINICAL TRIAL: NCT03575286
Title: Feasibility Study of an Automated Point-of-Care Urine Diagnostic Device for Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Voyant Diagnostics, Inc. (Industry)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Pregnancy Related
Keywords: Pregnancy; Urine Testing; Medical Diagnostics
MeSH Terms: interventions — Pregnancy Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- Pregnant female: Patient has been determined pregnant with a urine pregnancy test and, if applicable, a serum pregnancy test performed at Northwestern University.
  Interventions: Diagnostic Test: Pregnancy test
- Non-pregnant female: Patient has been determined not pregnant with a urine pregnancy test and, if applicable, a serum pregnancy test performed at Northwestern University.
  Interventions: Diagnostic Test: Pregnancy test

INTERVENTIONS:
Diagnostic Test: Pregnancy test — Detects hormone (hCG, Human Chorionic Gonadotropin) produced by the body during pregnancy

SUMMARY:
The primary purpose of this observational study is to demonstrate the feasibility of an automated point-of-care urine diagnostic device in determining the pregnancy status of patients through urine samples collected from patients at Northwestern University. Our hypothesis is that this automated point-of-care urine diagnostic device will be able to accurately determine a patient's pregnancy status at least 95% of the time.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18 years and older, upper age limit of 45 years
* Female patient
* Patients undergoing any procedures for pregnancy diagnosis and confirmation
* English speaking

The following special population will be included:

* Pregnant women

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, and teenagers)
* Prisoners

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female patients of childbearing age
Sampling Method: Non-Probability Sample
Enrollment: 123 (Estimated)
Dates: Start 2018-06-28 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Accuracy in determining pregnancy status | Time of collection - 1 month post collection
  Compare qualitative pregnancy test results generated by Voyant's device with urine pregnancy test result(s) and, if applicable, serum pregnancy test results performed at Northwestern University. From this comparison, we will determine the accuracy of Voyant's device. We will be using the same urine sample used at Northwestern.

CONTACTS AND LOCATIONS:
Overall Officials: MaryEllen Pavone, MD, MSCI, Principal Investigator — Northwestern University, Department of Obstetrics and Gynecology
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No